CLINICAL TRIAL: NCT05359302
Title: Effects of Ramadan Fasting on Sleeping and Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Chef of Emergency Deparment, University of Monastir
Other Study IDs: Sleeping and quality of life
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Fasting; Quality of Life; Sleep Disorder
Keywords: Ramadan Fasting; SF-36 score; sleeping score
MeSH Terms: conditions — Fasting; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Include participants who intend to practice Ramadan fasting and accept to complete the three part of the study .

DETAILED DESCRIPTION:
All volunteers and stable patients that intend to fast ramadan. Each participant is examined during three separate visits.

The week before Ramadan (Pre-R). the last week of Ramadan (R). the last week of the month following Ramadan (Post-R). Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patients clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.

All patients benifit of a routine examen and evaluation of the quality of life by Short Form 36 (SF36) test and sleeping by Pittsburg Sleep Quality Index (PQSI) score .

ELIGIBILITY:
Inclusion Criteria:

* Adult patient intending to fast Ramadan.

Exclusion Criteria:

* Age < 18 years old
* Hemodynamic instability.
* Myocardial infarction requiring urgent revascularization.
* Parkinsonism: tremor problem.
* Refusal, communication problem.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable patients that intend to fast Ramadan. Each participant is examined during three planned visits. The first takes place during the month preceding Ramadan. The second during the last week of Ramadan and the third thirty days after the end of Ramadan.
  Participants that miss one appointement or more are exluded from the study. Patient recrutement is conducted in primary care centers of the state of Monastir, out-patient clinic (Cardiology, Endocrinology) at the emergency department of Fattouma Bourguiba university hospital after a clarified written consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
the change in sleeping quality | the day of inclusion , 10 last day of Ramadan , 1 month after Ramadan
  the score of sleeping is calculated for each participant in the day of inclusion , then it is recalculated in the two others visits.
the change in the quality of life score | the day of inclusion , 10 last day of Ramadan , 1 month after Ramadan
  the score of quality of life is calculated for each participant in the day of inclusion , then it is recalculated in the two others visits.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Principal Investigator — University of Monastir
Locations (1):
- University hospital Fattouma Bourguiba, Monastir, Tunisia